CLINICAL TRIAL: NCT02331043
Title: Serum Cholesterol Reduction Efficacy of Biscuit With Added Plant Stanol Ester
Brief Title: Serum Cholesterol Reduction Efficacy of Biscuit With Plant Stanol Ester
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raisio Group (Industry)
Collaborators: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL 2012_034
Record Dates: First submitted 2014-12-31; First posted 2015-01-05 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Dyslipidemias; Hypercholesterolemia; Hyperlipidemias
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia; Hyperlipidemias | interventions — plant stanol ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo biscuit (Placebo Comparator): Biscuit without plant stanol ester
  Interventions: Dietary Supplement: Placebo
- Plant stanol ester biscuit (Experimental): Biscuit with plant stanol esters
  Interventions: Dietary Supplement: Plant stanol ester

INTERVENTIONS:
Dietary Supplement: Plant stanol ester
  Arms: Plant stanol ester biscuit
Dietary Supplement: Placebo
  Arms: Placebo biscuit

SUMMARY:
Efficacy of plant stanols as esters on LDL-cholesterol reduction is well documented. LDL-cholesterol lowering efficacy of the ingredient in a biscuit (providing 2 g plant stanols as esters per day) is less well known.

ELIGIBILITY:
Inclusion Criteria:

* mildly or elevated fasting serum cholesterol levels (between 5.2 to 6.5 mmol/l)
* fasting serum triglyceride levels below 3.0 mmol/l
* normal liver, kidney and thyroid function
* no lipid lowering medication
* no history of unstable coronary artery disease (myocardial infarction, coronary artery bypass craft (CABG), percutaneous transluminal coronary angioplasty (PTCA) within the previous 6 months, diabetes, temporal ischemic attack and malignant diseases

Exclusion Criteria:

* alcohol abuse (> 4 portion/per day)
* pregnancy
* use of plant stanol and plant sterol products and equivalent cholesterol lowering products, though the ones who have discontinued the consumption of these products minimum 3 weeks before the beginning of the study, can be included

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change (proportional) in LDL-c from baseline after 4-weeks' plant stanol ester biscuit consumption compared to controls | 4 weeks

SECONDARY OUTCOMES:
Change (proportional) in LDL-c from baseline after 4-weeks' plant stanol ester biscuit consumption in subjects consuming the biscuit with or without a meal | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wantanee Kriengsinyos, PhD, Principal Investigator — Mahidol University
Locations (1):
- Mahidon University, Nutrition Institute, Center of Innovation and Reference on Food for Nutrition (CIRFON), Phutthamonthon, Changwat Nakhon Pathom, Thailand